CLINICAL TRIAL: NCT00105144
Title: A Phase 3, Randomized, Double-Blind, Comparative Study of Micafungin (FK463) Versus Caspofungin as Antifungal Treatment in Patients With Invasive Candidiasis or Candidemia
Brief Title: Study of Micafungin in Patients With Invasive Candidiasis or Candidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-0-192; NCT00235742 (obsolete NCT alias)
Record Dates: First submitted 2005-03-07; First posted 2005-03-08 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Candidiasis; Candidemia
Keywords: Treatment Effectiveness; Treatment Efficacy; Investigational, Therapies; Antifungal, Systemic; Antibiotics, Antifungal; Micafungin
MeSH Terms: conditions — Candidiasis; Candidemia | interventions — Micafungin; Caspofungin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): lower dose
  Interventions: Drug: Micafungin
- 2 (Experimental): higher dose
  Interventions: Drug: Micafungin
- 3 (Active Comparator)
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Micafungin — IV
  Other Names: Mycamine; FK463
  Arms: 1; 2
Drug: Caspofungin — IV
  Other Names: Cancidas
  Arms: 3

SUMMARY:
The purpose of the study is to determine the safety and effectiveness of two dose levels of micafungin versus caspofungin in the treatment of proven invasive candidiasis or candidemia.

DETAILED DESCRIPTION:
The purpose of the study is to determine the efficacy and safety of two dose levels of micafungin versus caspofungin in the treatment of proven invasive candidiasis or candidemia. The maximum length of antifungal treatment is 4 weeks except in pre-defined patients where maximum length of therapy is 8 weeks. A post treatment assessment will be conducted at 2 weeks and 6 weeks after the last dose of all antifungal treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have candidemia or invasive candidiasis.

Exclusion Criteria:

* Patients who have received an echinocandin within one month prior to study entry.
* Patients who have received more than two days of prior systemic antifungal therapy for the current infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2004-09; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Overall treatment success, based on the investigator's assessment of pre-defined clinical and mycological response at the End of intravenous (IV) Therapy | End of therapy and 6 weeks post-treatment

SECONDARY OUTCOMES:
Overall treatment success, based on the Data Review Panel's assessment of pre-defined clinical and mycological response at the End of IV Therapy | End of therapy and 6 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (127):
- United States (52):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Los Angeles, California
  - San Francisco, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Bay Pines, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Maywood, Illinois
  - Beech Grove, Indiana
  - Evansville, Indiana
  - Des Moines, Iowa
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - St Louis, Missouri
  - Neptune City, New Jersey
  - Albany, New York
  - Manhasset, New York
  - New Hyde Park, New York
  - New York, New York
  - Rochester, New York
  - Stony Brook, New York
  - The Bronx, New York
  - Valhalla, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - West Reading, Pennsylvania
  - Providence, Rhode Island
  - Jackson, Tennessee
  - Memphis, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Fairfax, Virginia
  - Seattle, Washington
- Vienna, Austria
- Belgium (4):
  - Aalst
  - Brussels
  - Ghent
  - Liège
- Brazil (11):
  - Belo Horizonte, Mg-cep
  - Belo Horizonte, Minas Gerais
  - Cunitiba, Pr-cep
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Santos, São Paulo
  - São José do Rio Preto, São Paulo
  - São Paulo, São Paulo
  - Belo Horizonte
  - Salvador
  - São Paulo
- Canada (15):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Kingston, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Regina, Saskatchewan
  - Saskatoon, Saskatchewan
- Zagreb, Croatia
- Prague, Czechia
- France (5):
  - Bobigny
  - Metz
  - Paris
  - Strasbourg
  - Villejuif
- Germany (7):
  - Berlin
  - Bielefeld
  - Cologne
  - Frankfurt
  - Hanover
  - Ulm
  - Würzburg
- India (14):
  - Bangalore
  - Banglore
  - Chandigarh
  - Chennai
  - Cochin Kerala
  - Hyderabad
  - Kochi
  - Kolkotta
  - Lucknow
  - Ludhiana
  - Mangalore
  - Manipal
  - Mumbai
  - Uttar Pradesh
- Groningen, Netherlands
- Poland (3):
  - Gdansk
  - Lodz
  - Warsaw
- Spain (7):
  - Barakaldo
  - Barcelona
  - Madrid
  - Salamanca
  - Santander
  - Seville
  - Valencia
- Sankt Gallen, Switzerland
- United Kingdom (4):
  - London, England
  - Manchester, England
  - Glasgow, GB
  - Leeds, GB

REFERENCES:
- [Background] Pappas PG, Rotstein CM, Betts RF, Nucci M, Talwar D, De Waele JJ, Vazquez JA, Dupont BF, Horn DL, Ostrosky-Zeichner L, Reboli AC, Suh B, Digumarti R, Wu C, Kovanda LL, Arnold LJ, Buell DN. Micafungin versus caspofungin for treatment of candidemia and other forms of invasive candidiasis. Clin Infect Dis. 2007 Oct 1;45(7):883-93. doi: 10.1086/520980. Epub 2007 Aug 29. PMID 17806055
- [Derived] Shorr AF, Wu C, Kothari S. Outcomes with micafungin in patients with candidaemia or invasive candidiasis due to Candida glabrata and Candida krusei. J Antimicrob Chemother. 2011 Feb;66(2):375-80. doi: 10.1093/jac/dkq446. Epub 2010 Dec 8. PMID 21147825